CLINICAL TRIAL: NCT00664222
Title: Effects of Spironolactone on Insulin Resistance in Patients With Chronic Heart Failure
Brief Title: Spironolactone and Insulin Resistance in Chronic Heart Failure (CHF)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tottori University Hospital (Other)
Responsible Party: Kazuhide Ogino, MD, Center for Clinical Residency Program, Tottori University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: #344.1
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-04

CONDITIONS: Chronic Stable Heart Failure
Keywords: heart failure; insulin resistance; inflammatory cytokine; spironolactone; furosemide
MeSH Terms: conditions — Heart Failure; Insulin Resistance | interventions — Spironolactone; Furosemide

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: spironolactone + furosemide — spironolactone 25mg/day, 16 weeks and furosemide 20mg/day, 16weeks

SUMMARY:
The purpose of this study is to evaluate the effects of spironolactone and furosemide on insulin resistance in patients with chronic heart failure.

DETAILED DESCRIPTION:
Diuretics is useful in CHF patients. On the other hand, they deteriorate glucose metabolism. Therefore, the purpose of this study is to evaluate the effects of spironolactone and furosemide on insulin resistance in patients with chronic heart failure.

ELIGIBILITY:
Inclusion Criteria:

* chronic stable heart failure

Exclusion Criteria:

* renal dysfunction or under treatment with antidiabetic agents

Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2004-01; Study Completion 2005-12

PRIMARY OUTCOMES:
insulin resistance | 16 weeks